CLINICAL TRIAL: NCT05654649
Title: Dexamethasone in the Prevention of Post-spinal Paralytic Ileus After Cesarean Section, Does it Make a Difference: A Randomized Controlled Study
Brief Title: Dexamethasone in the Prevention of Post-spinal Paralytic Ileus After Cesarean Section
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: post-spinal paralytic ileus
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Ileus
MeSH Terms: interventions — Sodium Chloride; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Placebo Comparator): Patients received 5 ml of IV normal saline as a placebo just before spinal anesthesia
  Interventions: Drug: 0.9%sodium chloride
- Group D (Active Comparator): Patients received IV dexamethasone 8 mg in 5ml normal saline 0,9%, just before spinal anesthesia.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: 0.9%sodium chloride — Patients received 5 ml of IV normal saline as a placebo just before spinal anesthesia
  Arms: Group C
Drug: Dexamethasone — Patients received IV dexamethasone 8 mg in 5ml normal saline 0,9%, just before spinal anesthesia.
  Arms: Group D

SUMMARY:
Postoperative ileus is a perplexing problem for clinical surgeons. It occurs not only after abdominal surgery but also after any surgery that requires general anesthesia. Postoperative ileus is defined as the dysfunction of gastrointestinal motility after surgery, characterized by a decrease in, or stagnation of, intestinal peristalsis.

DETAILED DESCRIPTION:
Common clinical manifestations include abdominal pain, abdominal distention, nausea, vomiting, delayed flatus, delayed defecation, and inability to consume orally. Postoperative ileus is an uncomfortable experience, enhances the possibility of postoperative complications, prolongs hospital stay, and increases the economic burden. Postoperative gastrointestinal function recovery is of great concern. There is currently an urgent need to improve postoperative recovery of gastrointestinal function. The mechanism of Postoperative ileus varies, including autonomic regulation, inflammatory response, gastrointestinal hormones, and postoperative use of opioid drugs. Surgical gut damage destroys the intestinal barrier, stimulates the sympathetic and parasympathetic nervous systems, and enhances the release of inflammatory factors. These factors precipitate the occurrence of Postoperative ileus. The current use of laparoscopic techniques can reduce incision size and surgical trauma, enabling careful manipulation.

ELIGIBILITY:
Inclusion Criteria:

* •All participants will sign an informed consent prior to inclusion in the study.

  * All patients 18-40 years of full-term singleton pregnancy (37-41 weeks).,
  * American Society of Anaesthesiologists (ASA) classification class I and II scheduled.
  * for elective or semi-elective surgery (category 3 and 4 Caesarean sections).
  * All patients under spinal anesthesia for a Single baby pregnancy of more than 32 weeks will be included in this study.

Exclusion Criteria:

* will be patients' height < 150 or > 180 cm.
* Body mass index (BMI) >35 kg m-2.
* Contraindication or refusal to undergo regional anesthesia.
* any cardiovascular disease including arrhythmias and severe stenotic valvular heart disease.any renal or hepatic diseased patients.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
the time to first passage of flatus and or stool | 24 hours postoperative
  the time to first passage of flatus and or stool through the first 24 hours and the time of return of intestinal sounds,

CONTACTS AND LOCATIONS:
Locations (1):
- woman health hospital , Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Deng WW, Lan M, Peng AF, Chen T, Li ZQ, Liu ZL, Liu JM. The risk factors for postoperative ileus following posterior thoraco-lumbar spinal fusion surgery. Clin Neurol Neurosurg. 2019 Sep;184:105411. doi: 10.1016/j.clineuro.2019.105411. Epub 2019 Jul 1. PMID 31310924
- [Background] Petca A, Borislavschi A, Dumitrascu MC, Sandru F, Geoarsa M, Petca RC. Postoperative Ileus Complicated with Incomplete Evisceration after Hysterectomy for Benign Pathology. Chirurgia (Bucur). 2020 Jan-Feb;115(1):112-119. doi: 10.21614/chirurgia.115.1.112. PMID 32155406
- [Background] Holte K, Kehlet H. Postoperative ileus: a preventable event. Br J Surg. 2000 Nov;87(11):1480-93. doi: 10.1046/j.1365-2168.2000.01595.x. PMID 11091234
- [Background] Tevis SE, Carchman EH, Foley EF, Harms BA, Heise CP, Kennedy GD. Postoperative Ileus--More than Just Prolonged Length of Stay? J Gastrointest Surg. 2015 Sep;19(9):1684-90. doi: 10.1007/s11605-015-2877-1. Epub 2015 Jun 24. PMID 26105552